CLINICAL TRIAL: NCT02652325
Title: Comparison of Effectiveness of Povidone-iodine Versus Saline Versus 3M Skin and Nasal Antiseptic 5% Povidone-Iodine USP Swabs for Decolonizing Intranasal MSSA/MRSA
Brief Title: Nasal Swab studyComparison of Effectiveness of Povidone-iodine Versus Saline Versus 3M Skin and Nasal Antiseptic 5% Povidone-Iodine USP Swabs for Decolonizing Intranasal MSSA/MRSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016JPAR
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: MRSA/ MSSA Colonization of the Nares
MeSH Terms: interventions — Sodium Chloride; Povidone-Iodine

ARMS (3):
- povidone-iodine (Active Comparator)
  Interventions: Drug: Povidone-Iodine
- 3M Skin and Nasal Antiseptic 5% Povidone-Iodine USP swabs (Active Comparator)
  Interventions: Drug: 5% Povidone-Iodine USP swabs
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline
  Arms: Saline
Drug: Povidone-Iodine
  Arms: povidone-iodine
Drug: 5% Povidone-Iodine USP swabs
  Arms: 3M Skin and Nasal Antiseptic 5% Povidone-Iodine USP swabs

SUMMARY:
To determine if routinely available 10% povidone-iodine swabs are more effective than saline and 3M Skin and Nasal Antiseptic 5% Povidone-Iodine USP for decolonizing MRSA.

ELIGIBILITY:
Inclusion Criteria:

1. All potential total hip and total knee arthroplasty candidates
2. All femoroacetabular osteoplasty patients
3. All pelvic acetabular osteotomy patients
4. All core decompression patients

Exclusion Criteria:

1. Any trauma patients
2. Any tumor patients
3. Any patient with periprosthetic joint infection
4. Any patient with surgical site infection
5. Any patient with known MRSA infection
6. Any patients allergic to povidone-iodine
7. Patients with thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
MSSA/MRSA colonization in the nares | 4 hours
  Subjects will undergo a swab of their nares to undergo PCR analysis to determine if they are effectively decolonized four hours after initial treatment
MSSA/MRSA colonization as tested by PCR | 24 hours
  Subjects will undergo a swab of their nares to undergo PCR analysis to determine if they are effectively decolonized four hours after initial treatment

REFERENCES:
- [Derived] Rezapoor M, Nicholson T, Tabatabaee RM, Chen AF, Maltenfort MG, Parvizi J. Povidone-Iodine-Based Solutions for Decolonization of Nasal Staphylococcus aureus: A Randomized, Prospective, Placebo-Controlled Study. J Arthroplasty. 2017 Sep;32(9):2815-2819. doi: 10.1016/j.arth.2017.04.039. Epub 2017 May 3. PMID 28578841